CLINICAL TRIAL: NCT00935064
Title: Effect of Renin Inhibition on Cardiovascular Autonomic Nerve Function in Diabetes
Brief Title: The Effect of Renin Inhibition on Nerve Function in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29011; NIH (INBRE 2-P20-RR016472-09)
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Results first posted 2013-04-01 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Active Comparator): Pill, 300 mg, once daily, for 6 weeks
  Interventions: Drug: Aliskiren; Other: Placebo
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aliskiren — Pill, 300 mg, once daily, for 6 weeks
  Arms: Aliskiren
Other: Placebo — Placebo orally one tablet once a day for 6 weeks.

SUMMARY:
This study will assess the effect of direct renin inhibition on nerve function in persons with diabetes using a double-blind, placebo-controlled randomized trial involving two treatment arms (i.e., [1] 30 participants enrolled and randomized to 300 mg of Aliskiren; [2] 30 participants enrolled and randomized to placebo).

ELIGIBILITY:
Inclusion Criteria:

* Individuals >18 years old with type 1 or type 2 diabetes mellitus.

Exclusion Criteria:

* Individuals currently taking the maximum dose of an ACE inhibitor or an ARB.
* Individuals with a history of a MI, percutaneous coronary interventions, coronary artery bypass graft (CABG) surgery, acute coronary syndromes, recent/on going atrial fibrillation, frequent atrial arrhythmias, frequent ventricular arrhythmias, or acute myocardial ischemia changes.
* Individuals whose treatment dosage changes 2 months prior to the study for antihypertensive and antidiabetes medications, and the following medications that may affect the ANS: anti-tuberculosis drugs, nitrofurantoin, metronidazole, chloramphenicol, perhexiline maleate, amiodarone, clofibrate, tricyclic antidepressants, phenytoin, barbiturates, neuroleptic, antiparkinsonism drugs, and nitrated drugs.
* Pregnant or lactating females.
* Individuals with impaired renal function (i.e., creatinine >1.5 mg/dl), a history of dialysis, nephritic syndrome or renovascular hypertension.
* Individuals with potassium levels within 0.5 mmol/L of the upper limit of normal (i.e., hyperkalemia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raelene E Maser, PhD, Principal Investigator — University of Delaware
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren: 300 mg, once daily, for 6 weeks
- Placebo: Once daily, for 6 weeks
Period: Overall Study
Arm/Group | Aliskiren | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 26 | 55
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12) | 53 (12) | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 14 | 19 | 33
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure Before and After Treatment
Description: Systolic blood pressure at baseline and follow-up
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 30 | 30
mm Hg
  Baseline | 121.0 (11.3) | 124.1 (13.8)
  Follow-up | 112.1 (12.1) | 121.5 (15.2)

2. Primary Outcome: Diastolic Blood Pressure Before and After Treatment
Description: Diastolic blood pressure at baseline and follow-up.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 30 | 30
mm Hg
  Baseline | 66.1 (7.0) | 68.2 (8.3)
  Follow-up | 61.5 (6.5) | 66.7 (9.3)

3. Primary Outcome: Serum Renin Level Before and After Treatment
Description: Serum renin level at baseline and follow-up
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: ug/l/h
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 30 | 30
ug/l/h
  Baseline | 2.4 (3.8) | 3.1 (6.0)
  Follow-up | 0.5 (0.4) | 2.6 (4.2)

4. Primary Outcome: Mean Circular Resultant Before and After Treatment
Description: Mean circular resultant at baseline and follow-up. There are several different assessment modalities used for the determination of cardiovascular autonomic function (i.e. HRV). One widely used clinical method for assessing HRV is RR-variation during deep breathing. RR-variation is a measure of the change in heart rate resulting from the variation in intrathoracic pressure due to respiration. It is predominantly a function of parasympathetic activity. In this study, RR-variation during deep breathing, performed for 6 min, was measured by vector analysis [i.e. mean circular resultant (MCR)] and by the expiration/inspiration (E/I) ratio of the first six breath cycles. With regard to the MCR, the length of the vector mean is proportional to the degree of HRV. Weinberg and Pfeifer first introduced the assessment of HRV via determination of the MCR in a paper in Biometrics 1984:40:855-861. Low HRV is considered to be less favorable.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: MCR is unitless
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 30 | 30
MCR is unitless
  Baseline | 41.8 (19.7) | 38.2 (23.6)
  Follow-up | 50.8 (26.1) | 37.5 (24.1)

5. Primary Outcome: Expiration/Inspiration Ratio Before and After Treatment
Description: Expiration/inspiration ratio at baseline and follow-up. There are several different assessment modalities used for the determination of cardiovascular autonomic function (i.e. HRV). One widely used clinical method for assessing HRV is RR-variation during deep breathing. RR-variation is a measure of the change in heart rate resulting from the variation in intrathoracic pressure due to respiration. It is predominantly a function of parasympathetic activity. In this study, RR-variation during deep breathing, performed for 6 min, was measured by vector analysis [i.e. mean circular resultant (MCR)] and by the expiration/inspiration (E/I) ratio of the first six breath cycles.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 30 | 30
Ratio
  Baseline | 1.22 (0.12) | 1.21 (0.14)
  Follow-up | 1.28 (0.15) | 1.20 (0.14)

ADVERSE EVENTS:
Arm/Group | Aliskiren | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 3/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aliskiren (N=30) | Placebo (N=30)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No